CLINICAL TRIAL: NCT04931550
Title: Clinical Study of Impact of Different Pacing Site in Patients
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: Y2020-675
Record Dates: First submitted 2021-06-14; First posted 2021-06-18 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Bradyarrhythmias; Heart Failure; Pacemaker
MeSH Terms: conditions — Bradycardia; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pacemaker implantation — Different pacing sites will be chosen according to the patients condition.

SUMMARY:
At present, cardiac pacing has been widely used in the treatment of bradyarrhythmias and heart failure, which can effectively improve the survival rate of patients. With the rapid development of technology, different sites can be chosen to pace, such as right atrial appendage, the atrial septum and the right atrial wall in the atrium, His bundle, left bundle branch area, right ventricular apex, outflow tract, and left ventricular pacing via coronary vein in the ventricle. There are few studies comparing the long-term efficacy and safety of different pacing sites in daily practice. This study aims to observe the efficacy and safety of cardiac pacing at different sites in short and long term, and to compare the advantages and disadvantages of pacing at different sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received pacemaker implantation in the Second Hospital of Zhejiang Medical University by Pan Xiaohong and other surgeons.
* Patients who have the ability to understand the test and can cooperate with investigators.

Exclusion Criteria:

* Patients who unable to understand or unwilling to fill in informed consent forms or follow visitors.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the current reports and the researcher's pacing implantation status, with an enrollment rate of 90% and a loss of follow-up rate of 10%, it is estimated that 600 cases were screened, 540 cases were selected, and about 500 cases were effective.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Composite of Cardiovascular death, myocardial infarction, and stroke events | 60 months
  Composite of Cardiovascular death, myocardial infarction, and stroke events in 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China